CLINICAL TRIAL: NCT06024980
Title: Department of Otolaryngology Head Neck Surg
Brief Title: Using the Subglottic Pressure to Predict the Dysphagia After Partial Laryngectomy
Acronym: SPPDPL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-59
Record Dates: First submitted 2023-08-21; First posted 2023-09-06 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Laryngeal Cancer; Dysphagia
Keywords: partial laryngectomy; subglottic pressure; laser
MeSH Terms: conditions — Laryngeal Neoplasms; Deglutition Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supraglottic and glottic T2 laryngeal carcinoma (Active Comparator): The open partial horizontal laryngectomy was underwent in patients with supraglottic or glottic laryngeal carcinoma in T2
  Interventions: Procedure: Open partial horizontal laryngectomy(OPHL), Type I-III
- Supraglottic and glottic T1 laryngeal carcinoma (Active Comparator): The transoral endoscopic laser cordectomy was underwent in patients with supraglottic or glottic laryngeal carcinoma in T1
  Interventions: Procedure: Transoral endoscopic laser cordectomy

INTERVENTIONS:
Procedure: Open partial horizontal laryngectomy(OPHL), Type I-III — An open partial horizontal laryngectomy(OPHL) was performed for patients with T2 supraglottic and glottic carcinoma, according to the American Joint Committee on Cancer(AJCC) criteria. Type I OPHL: Entails the resection of the supraglottis, including the pre-epiglottic space and the upper half of the thyroid cartilage. Type II OPHL: Entails the resection of the entire thyroid cartilage, with the inferior limit represented by the upper edge of the cricoid ring. Type III OPHL: Entails the resection of the entire supraglottic, glottic, and part of the subglottic sites, sparing both or at least one functioning crico-arytenoid unit.
  Other Names: Type I OPHLs(formerly defined horizontal supraglottic laryngectomy), Type II (previously called supracricoid laryngectomy), and Type III (also named supratracheal laryngectomy).
  Arms: Supraglottic and glottic T2 laryngeal carcinoma
Procedure: Transoral endoscopic laser cordectomy — For patients with T1 glottic laryngeal carcinoma, according to the criteria of the American Joint Committee on Cancer(AJCC), transoral endoscopic CO2 laser(2-40Watts) cordectomy was performed. The classification comprises eight types of cordectomies:
  * A subepithelial cordectomy (type I) is a resection of the epithelium of the vocal fold.
  * A subligamental cordectomy (type II) is a resection of the epithelium, Reinke's space, and vocal ligament.
  * Transmuscular cordectomy (type III), which proceeds through the vocalis muscle.
  * Total cordectomy (type IV).
  * Extended cordectomy encompasses the contralateral vocal fold and the anterior commissure (type Va).
  * Extended cordectomy, which includes the arytenoid (type Vb).
  * Extended cordectomy, which encompasses the subglottis (type Vc).
  * Extended cordectomy, which consists of the ventricle (type Vd).
  Other Names: Transoral carbon dioxide(CO2) laser microsurgery
  Arms: Supraglottic and glottic T1 laryngeal carcinoma

SUMMARY:
Recruited patients are divided into two arms depending on laryngeal carcinoma's T1 and T2 stages. Two interventions were undergone, including transoral endoscopic laser cordectomy and open partial horizontal laryngectomy (OPHL). During the pre-and post-operative time, patients performed measurements of swallowing function, including direct subglottic pressure, Eating Assessment Tool-10(EAT-10) questionnaire, swallowing ability to different textures, and fiberoptic evaluation of swallowing(FEES). Patients undergo subglottic pressure measurement and swallowing function evaluation three times: 3-7 days, two months, and six months after surgery. Patients also performed measurement voice acoustic analysis and subjective assessment one-day pre-operation and six months post-operation.

DETAILED DESCRIPTION:
There were swallowing disorders after partial laryngectomy in most patients with laryngeal carcinoma. At least these patients need several months to recover. Few people required surgery of total laryngectomy to maintain normal swallowing function. The swallowing training cannot acquire a valid swallowing function and take the risk of aspiration pneumonia. Factors that influenced the swallowing function recovery, for example, the time of nasogastric feeding and tracheostomy tube removal, were affected by age and diabetes.

On the other hand, the pharynx size of a CT scan can predict the recovery of swallowing function after laryngectomy. But those are not directly related to swallowing motion, although they are predictors of dysphagia. The investigators will perform the study with swallowing function measures to find predictors relative to swallowing function and evaluate dysphagia's recovery early.

Subglottic pressure is a protective factor that can reduce aspiration risk. This research will measure the subglottic pressure after laryngectomy and predict or monitor swallowing disorders. Specific objectives were to verify the effect of laryngectomy on subglottic pressure.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80 years
* Surgical treatment by open partial horizontal laryngectomy type I or II and transoral laser cordectomy for squamous cell carcinoma
* Availability of clinical data
* Validity of normal swallowing of thin liquids

Exclusion Criteria:

* Presence of severe chronic obstructive pulmonary disease, severe heart disease, and psychopathy or mental disease
* Surgery complications(such as sepsis, pharyngocutaneous fistula, surgical revision)
* Radiotherapy histology
* Swallowing disorder or trachea aspiration before surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Fiberoptic laryngoscope evaluation of swallowing | Pre-operation, one week post-operation, two months post-operation, six months post-operation
  The patient, in a sitting position, had to swallow liquid. The tip of a flexible endoscope was positioned beyond the soft palate, and the pharyngeal phase of swallowing was studied, recording videos and images for further analysis. In particular, according to the severity scale, the scores ranged from 1 point (no materials entered the airway) to 8 points (the material penetrated below the vocal cords, but no effort was made to eject the material), representing the severity of risk for penetration
direct subglottic pressure | At one day before surgery, one week after surgery, two months after surgery, six months after surgery
  Subglottic pressure was measured while swallowing a thinned solution with and without airflow delivery through the subglottic puncture needle. The unit of subglottic pressure is cmH20.
EAT-10 questionnaire | At one day before surgery, two months after surgery, six months after surgery
  The EAT-10 questionnaire consists of a 10-item questionnaire with a maximum total score of 40 points. All items are rated on a 5-point scale in which 0 indicates no problem, and 4 indicates a severe problem in swallowing function. An EAT-10 score of over 3 is abnormal and indicates a higher self-perception of the presence of dysphagia.
Swallowing ability to four different textures | At one day before surgery, one week after surgery, two months after surgery, six months after surgery
  An early 5-point scoring system (score one corresponding to the early postoperative assessment) was applied to each patient depending on his ability to swallow one to four different textures (liquid, semi-liquid, semi-solid, and solid). A score of 0 is poor (no power to swallow), while a score of 4 is good.

SECONDARY OUTCOMES:
Voice acoustic analysis | At one day before surgery, six months after surgery
  Every participant was asked to phonate a sustained vowel /a/ at a habitual comfortable pitch and intensity for voice pitch, quality assessments, and habitual vocal intensity. The recordings were made in a quiet clinical room. The participant sat in front of a microphone positioned approximately 10cm from the left corner of the mouth. The voice signal coupled with Roland's Audio interface with a sampling rate of 44k-Hz and 16-bit accuracy. The signal was stored in a computer system after collecting sustained vowels. The voice signals were analyzed using speech analysis software. The stable phase of the voice sample was extracted for analysis. The 3,000-msec sample was analyzed for acoustic parameters. The voice acoustic parameters include F0 (fundamental frequency) in Hertz(Hz), percentage of jitter(%), percentage of shimmer(%), Harmonic to noise ratio(HNR), and intensity in decibels(dB).
The time in weeks of nasogastric feeding | At two months after surgery, six months after surgery
  The duration of surgery to oral feeding after withdrawing naso tube.

CONTACTS AND LOCATIONS:
Overall Officials: Xujiao Chen, Ms, Principal Investigator — Guangdong Provicial People's Hospital（Guangdong Academy of Sciences), Southern Medical University
Locations (1):
- Guangdong Provincial People's hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bagwell K, Leder SB, Sasaki CT. Is partial laryngectomy safe forever? Am J Otolaryngol. 2015 May-Jun;36(3):437-41. doi: 10.1016/j.amjoto.2014.11.005. Epub 2014 Nov 20. PMID 25595047
- [Background] Freitas AS, Santos IC, Furia C, Dornelas R, Silva ACAE, Dias FL, Salles GF. Prevalence and associated factors of aspiration and severe dysphagia in asymptomatic patients in the late period after open partial laryngectomy: a videofluoroscopic evaluation. Eur Arch Otorhinolaryngol. 2022 Jul;279(7):3695-3703. doi: 10.1007/s00405-021-07231-4. Epub 2022 Jan 4. PMID 34982204
- [Background] Breunig C, Benter P, Seidl RO, Coordes A. Predictable swallowing function after open horizontal supraglottic partial laryngectomy. Auris Nasus Larynx. 2016 Dec;43(6):658-65. doi: 10.1016/j.anl.2016.01.003. Epub 2016 Feb 4. PMID 26853312
- [Background] Dawson C, Pracy P, Patterson J, Paleri V. Rehabilitation following open partial laryngeal surgery: key issues and recommendations from the UK evidence based meeting on laryngeal cancer. J Laryngol Otol. 2019 Mar;133(3):177-182. doi: 10.1017/S0022215119000483. PMID 30983563
- [Background] Clarett M, Andreu MF, Salvati IG, Donnianni MC, Montes GS, Rodriguez MG. [Effect of subglottic air insufflation on subglottic pressure during swallowing]. Med Intensiva. 2014 Apr;38(3):133-9. doi: 10.1016/j.medin.2013.01.003. Epub 2013 Mar 6. Spanish. PMID 23473519
- [Background] Alaskarov E, Ozturk O, Batioglu-Karaaltin A, Gulmez ZD, Erdur ZB, Inan HC. Functional Outcomes of the Hyaluronic Acid Injections in Patients Who Underwent Partial Laryngectomy. J Voice. 2022 May;36(3):417-422. doi: 10.1016/j.jvoice.2020.06.026. Epub 2020 Jul 22. PMID 32712078
- [Background] Fakhry N, Michel J, Giorgi R, Robert D, Lagier A, Santini L, Moreddu E, Puymerail L, Adalian P, Dessi P, Giovanni A. Analysis of swallowing after partial frontolateral laryngectomy with epiglottic reconstruction for glottic cancer. Eur Arch Otorhinolaryngol. 2014 Jul;271(7):2013-20. doi: 10.1007/s00405-013-2750-3. Epub 2013 Oct 8. PMID 24100885